CLINICAL TRIAL: NCT00023088
Title: Rehabilitation Medicine Screening Protocol
Brief Title: Screening Study for the Department of Rehabilitation Medicine
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940130; 94-CC-0130
Record Dates: First submitted 2001-08-22; First posted 2001-08-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-09

CONDITIONS: Convalescence; Healthy
Keywords: Rehabilitation; Functional Level; Activity of Daily Living; Mobility; Normal Volunteer
MeSH Terms: conditions — Convalescence

SUMMARY:
The primary function of the Department of Rehabilitation Medicine (RMD) is to diagnose and treat patients at the NIH who have problems in locomotion, activities of daily living, occupational roles, communication, swallowing, or problems with chronic pain. The major goal of this department s to help patients achieve maximal function so that they can resume their daily living activities as normal as possible.

In order for the department to accomplish it's goal it requires the involvement of medical staff and the use of a variety of tests and instruments. Before a new test, evaluation technique, or piece of physical equipment can be considered for use in the treatment of patients it must be carefully studied.

Researchers must make sure the test, technique, or instrument is safe, sensitive, accurate, specific, and reproducible. Therefore all of these tests, techniques, and instruments must first undergo a trial period. Normal volunteers and patients from the RMD and outside of the RMD may be selected to participate in the trial period.

This study provides a framework for researchers in the Department of Rehabilitation Medicine (RMD) to develop new tests, techniques, technology, and equipment.

DETAILED DESCRIPTION:
This protocol provides a framework for clinicians in the Department of Rehabilitation Medicine (RMD) to develop and pilot new tests, techniques, technology, or equipment to remain state-of-the-art.

ELIGIBILITY:
* INCLUSION CRITERIA:

In- and outpatients referred to the Rehabilitation Medicine Department.

Normal volunteers of either sex.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1994-04-13; Study Completion 2008-07-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States